CLINICAL TRIAL: NCT00101985
Title: An Eight-week, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate Efficacy and Safety of Talnetant in Subjects With Irritable Bowel Syndrome
Brief Title: Eight-Weeks Of Treatment With Talnetant In Subjects With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 223412/068
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Colon
Keywords: Quality of Life; Irritable bowel syndrome; IBS; SB223412; Qol
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — SB 223412

INTERVENTIONS:
Drug: talnetant

SUMMARY:
This study will evaluate the effectiveness and safety of the investigational drug talnetant in treating subjects with irritable bowel syndrome (IBS).

ELIGIBILITY:
Inclusion criteria:

* Subjects will be required to conduct self-assessments of their IBS symptoms using a touch-tone telephone system for the duration of the study (15 weeks).
* Must be diagnosed with IBS consistent with the Rome II criteria.
* Must have normal results from a colonic procedure within 2 years of randomization.
* Must have conducted self-assessments on at least 12 days and have a documented average IBS pain or discomfort score of greater than or equal to 1.5 during the two-week screening phase.

Exclusion criteria:

* Self-assessment of no stool for 7 days during the two-week screening phase.
* Clinically significant abnormal laboratory tests.
* Current evidence or history of various conditions, comorbidities, or surgeries such as Irritable Bowel Disease (IBD), gastrointestinal surgeries, and diverticulitis.
* Inability to use the touch-tone telephone system.
* Hypersensitivity to quinolone antibiotics or quinolone derivatives.
* Diagnosis of a psychiatric disorder within the past 2 years and not on a stable dose of medication for at least 6 months.
* Women who are pregnant, breast feeding, or planning to become pregnant during the study.

Permitted medications: The subject is allowed to take any of the following medications, provided they maintain a stable dose for at least 30 days prior to the Screening visit and throughout the remainder of the study:

* Antidepressants, except REMERON
* Antihypercholesterolemics
* Iron supplements
* Bulking agents
* Fiber supplement
* Thyroid replacement therapy (levothyroxine)
* Antipsychotics
* Cox-2 inhibitors (CELEBREX)

Prohibited medications: Subjects must stop taking any medications they are taking to treat their IBS symptoms and must not have taken any of the prohibited medications at least 7 days prior to the Screening visit and must remain off these medications for the duration of the study.

* Anticholinergics (dicyclomine, hyoscyamine, propantheline)
* Cholinomimetic (bethanechol, pyridostigmine, tacrine, physostigmine)
* All narcotics (morphine, codeine, TYLENOL #3, propoxyphene, either alone or in combination)
* Tramadol hydrochloride (ULTRAM)
* Colchicine
* Orlistat (XENICAL)
* Misoprostol, alone or in combination (ARTHROTEC, CYTOTEC)
* 5-HT3 receptor antagonists (ondansetron, tropisetron, dolasetron, granisetron, mirtazapine, cilansetron, alosetron)
* Tegaserod (ZELNORM)
* Gabapentin
* Lupron
* Antacids containing magnesium or aluminium
* Antidiarrheal agents
* Bismuth compounds
* Prokinetic agents (cisapride, metoclopramide)
* Sulfasalazine
* Laxatives
* Cholestyramine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2004-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Determine whether talnetant provided adequate relief from IBS pain and discomfort for at least one of three talnetant dose groups compared with placebo and to determine the safety and tolerability of talnetant in subjects with IBS.

SECONDARY OUTCOMES:
- Explore response among subgroups IBS. - Evaluate positive treatment effects within bowel subgroups. - Compare treatment groups for global improvement of IBS symptoms. - Improvement of IBS pain or discomfort, Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (122):
- United States (66):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Bristol, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Torrington, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Riverside, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Florence, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Salisbury, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Blackwood, New Jersey
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Fishkill, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Newtown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Lacey, Washington
- Australia (12):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Newtown, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Spring Hill, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Port Lincoln, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Malvern, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Canada (13):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- France (8):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Issoire
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Miramas
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Vitry-sur-Seine
- Germany (6):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Stadskanaal, Netherlands
- South Africa (4):
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, N1 City
  - GSK Investigational Site, Parktown
  - GSK Investigational Site, Somerset West
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Oviedo
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Nacka
  - GSK Investigational Site, Stockholm
- United Kingdom (4):
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Portergate, Sheffield
- GSK Investigational Site